CLINICAL TRIAL: NCT06615596
Title: Discontinuation of Anticoagulations After Successful Catheter Ablation of Atrial Fibrillation: DESTINATION Study
Brief Title: Discontinuation of Anticoagulations After Successful Catheter Ablation of Atrial Fibrillation
Acronym: DESTINATION
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Yan Yao, MD,PhD, Director, Arrhythmia Center, Fu Wai Hospital, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCRCSZ-2023-011
Record Dates: First submitted 2024-09-22; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Catheter Ablation; Anticoagulation Discontinuation; Post-Ablation Monitoring; Randomized Controlled Trial; Thromboembolic Risk; Smart Wearable Devices; AF Recurrence Detection
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anticoagulants; Catheter Ablation

STUDY DESIGN:
Intervention Model Description: The intervention in this study involves two arms: patients either continue or discontinue anticoagulation therapy after successful catheter ablation for atrial fibrillation (AF). Participants in the continuation arm will receive non-vitamin K antagonist oral anticoagulants (NOACs) such as dabigatran, rivaroxaban, apixaban, etc or warfarin tailored to their specific risk profiles. The discontinuation arm will cease anticoagulation therapy following randomization. Smart wearable devices will monitor for AF recurrence, and patients will be followed for 24 months, with primary endpoints including thromboembolic and bleeding events.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- on-OAC (Active Comparator): In the cohort assigned to the "on-OAC" arm, which entails the continuation of Oral Anticoagulant (OAC) therapy, patients were prescribed Non-Vitamin K Antagonist Oral Anticoagulants (NOACs), specifically dabigatran, rivaroxaban, or apixaban, for a duration of 24 months following randomization. The dosing regimen was as follows: (1) Standard dosage included rivaroxaban at 20mg daily, apixaban at 5mg twice daily, and dabigatran at 150mg twice daily. (2) Reduced dosage was administered in cases where patients were aged over 75 years, had a body weight less than 50kg, or exhibited creatinine clearance below 50ml/min.
  Interventions: Drug: Anticoagulant drugs; Procedure: Catheter Ablation
- off-OAC (Experimental): In the off-OAC, involving the discontinuation of OAC therapy, patients had their OAC treatment terminated post-randomization, and no placebo medication was administered as a substitute.
  Interventions: Behavioral: discontinue anticoagulation therapy; Procedure: Catheter Ablation

INTERVENTIONS:
Behavioral: discontinue anticoagulation therapy — Participants in the discontinuation arm will cease anticoagulation therapy following randomization. Smart wearable devices will monitor for AF recurrence, and patients will be followed for 24 months, with primary endpoints including thromboembolic and bleeding events.
  Arms: off-OAC
Drug: Anticoagulant drugs — Participants in the continuation arm will receive oral anticoagulant drugs such as dabigatran, rivaroxaban, apixaban, warfarin, etc. tailored to their specific risk profiles. The discontinuation arm will cease anticoagulation therapy following randomization. Smart wearable devices will monitor for AF recurrence, and patients will be followed for 24 months, with primary endpoints including thromboembolic and bleeding events.
  Arms: on-OAC
Procedure: Catheter Ablation — Catheter ablation is a medical procedure used to treat atrial fibrillation (AF) by targeting and destroying small areas of heart tissue that cause irregular heartbeats. Using a specialized catheter, radiofrequency energy, cryotherapy, or pulsed field ablation (PFA) is applied to isolate the pulmonary veins or ablate other specific heart areas. The goal is to restore normal heart rhythm by electrically isolating problematic areas responsible for AF. This FDA-regulated procedure is minimally invasive and requires follow-up monitoring for AF recurrence and other potential complications. No specific ablation technique is mandated, allowing flexibility for operators to choose based on their expertise and center practices. The ablation strategy may include pulmonary vein isolation or additional procedures based on the type of AF. This approach distinguishes the study by providing real-world applicability, reflecting the diversity of ablation methods used in clinical practice.

SUMMARY:
The DESTINATION Study investigates whether anticoagulation therapy is necessary after successful catheter ablation (CA) for atrial fibrillation (AF). Current guidelines recommend continued anticoagulation based on stroke risk scores, even post-ablation, potentially exposing patients to unnecessary bleeding risks. This international, multicenter, randomized controlled trial aims to compare thromboembolic and bleeding event risks between patients who continue and discontinue anticoagulation after ablation. The study involves 3,160 AF patients, all free of AF recurrence within 6 months to 1 year after ablation. Smart wearable monitors will track recurrence, and patients are followed for 24 months to assess event rates. Findings may reshape anticoagulation guidelines, improving clinical practice for AF patients worldwide.

DETAILED DESCRIPTION:
This prospective, international, multicenter randomized controlled trial (RCT) investigates the safety and necessity of continuing anticoagulation therapy after successful catheter ablation of atrial fibrillation. The study will enroll 3,160 patients who underwent catheter ablation for AF and achieved no recurrence within 6 months to 1 year post-procedure. Participants will be randomly assigned to either continue or discontinue anticoagulation therapy. Smart wearable devices will monitor AF recurrence every 3 months, detecting both symptomatic and asymptomatic events. The study's primary endpoint is a composite of ischemic stroke, systemic embolism, and major bleeding at a 24-month follow-up. Secondary outcomes include AF recurrence rates, re-ablation needs, and quality of life measures. Participants are monitored through follow-up visits at 3, 6, 12, 18, and 24 months, and data from wearable devices will be transmitted to the research team. This study is significant due to the diversity of the population, with sites in China and the US, allowing for results that are generalizable across ethnic and geographic lines. The trial's findings aim to provide high-quality evidence to inform future guideline recommendations regarding post-ablation anticoagulation therapy, potentially reducing unnecessary bleeding risks and optimizing treatment outcomes. The inclusion of smart wearable monitors enhances the detection of asymptomatic recurrences and provides continuous, reliable data on patient health during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosed paroxysmal, persistent, or longstanding persistent AF
* Successful procedure (defined as restoration of sinus rhythm after PV isolation for paroxysmal AF, restoration of sinus rhythm after PV isolation and completion of additional ablation for persistent AF, according to 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation) and no recurrence within 3 months of ablation, using a cooled tip RF-, laser- or cryo-balloon-catheter
* No periprocedural complications
* Signed informed consent
* Male with CHA2DS2-VASC score ≥1, female with score ≥2.

Exclusion Criteria:

* Valvular AF (moderate- severe mitral insufficiency; relevant mitral stenosis with a mean pressure gradient >5mmHg)
* Reversible AF (e.g. uncontrolled hyperthyroidism)
* Prior AF ablation (including surgical ablation)
* History of left atrial appendage occlusion/ligation/excision
* Concomitant surgical ablation
* Left atrial diameter >50 mm
* Left atrial or LAA thrombus
* Pregnancy/breast feeding
* Women of childbearing age who refuse to use a highly effective and medically acceptable form of contraception throughout the study
* Patient has a non-arrhythmic condition necessitating long-term oral anticoagulation (i.e. PE, ventricular thrombus, peripheral thrombosis, etc)
* Recent myocardial infarction, NYHA class IV heart failure, patent foramen ovale, recent trauma or other prothrombotic conditions
* Patient with special risk factors for stroke unrelated to AF, specifically known thrombophilia/ hypercoagulability, uncontrolled hypertension (systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg within 4 days of enrollment), untreated familial hyperlipidemia, known vascular anomaly (intracranial aneurysm/ arteriovenous malformation or chronic vascular dissection), or known severe carotid disease.
* Patient has bleeding contra-indication to oral anticoagulation (such as bleeding diathesis, hemorrhagic disorder, significant gastrointestinal bleeding within 6 months, intracranial/intraocular/ atraumatic bleeding history, fibrinolysis within 48 hours of enrollment).
* Patient has other contraindication to oral anticoagulation or treatment with antiplatelet agent
* Patient has been on strong CYP3A inducers (such as rifampicin, phenytoin, phenobarbital, or carbamazepine) or strong CYP3A inhibitors (such as ketoconazole or protease inhibitors) within 4 days of enrolment
* Structural congenital heart disease
* Recent stroke or intracranial hemorrhage within 6 months
* Inability to adequately understand nature, significance, implications and risks of study precipitation and to comply with follow-up (i.e. bipolar disorders, severe depression, suicidal tendencies, among others) as judged by the local physician, ongoing drug or alcohol addiction (> 8 drinks/week)
* Patients who are > 85 years of age
* Patients who are critically ill or who have a life expectancy <3 years
* Patient is unable or unwilling to provide informed consent
* Patient is included in another randomized clinical trial or a clinical trial requiring an insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3160 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Composite outcome consisting of thromboembolic events and clinically significant bleeding events | 24 month
  The primary endpoint of this study comprises a composite outcome consisting of thromboembolic events and clinically significant bleeding events. Specifically, it encompasses the following components:
  1. Incidence of ischemic stroke and systemic thromboembolism within the 2-year post-ablation period in each respective study group.
  2. Incidence of clinically significant bleeding within the 2-year post-ablation period in each respective study group.
  Unit of Measure: Number of events (strokes, systemic embolism, major bleeding episodes).

SECONDARY OUTCOMES:
AF Recurrence Rate | 24 month
  Percentage of patients with documented AF recurrence at 2 years.
Repeat Ablation Proportion | 24 month
  Percentage of patients undergoing repeat ablation within each group
Thromboembolic/Bleeding Event Rates after repeat procedure | 24 month
  Percentage of patients with Thromboembolic and Bleeding events after repeat ablation in each group
Thromboembolic/Bleeding Event Rates after recurrence in off-OAC | 24 month
  Percentage of patients with thromboembolic and bleeding event rates in patients resuming anticoagulation therapy due to AF recurrence in the no anticoagulation group
Major Adverse Cardiovascular Events (MACE) | 24 month
  Number of MACE events including acute coronary syndrome, acute myocardial infarction (MI), serious arrhythmias, heart failure, cardiovascular mortality, and all-cause mortality in each group
Complication rates | 24 month
  Incidence rates of complications include bleeding, cardiac tamponade, vascular damage, pulmonary vein stenosis, stroke or thromboembolism, heart block, esophageal injury, infection, etc. based on different ablation method

CONTACTS AND LOCATIONS:
Locations (12):
- Brigham and Women Hospital, Boston, Massachusetts, United States
- China (11):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen, Guangdong
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cardiovascular Hospital (Shanxi Cardiovascular Research Institute), Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Yunnan Fuwai Cardiovascular Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No